CLINICAL TRIAL: NCT06377306
Title: Identifying Periods of High Training Load Considering the Menstrual Cycle Phases in Elite and Non-elite Female Athletes Using Measures of Strength, Fatigue, Injury, Psychological Parameters, Serum Circulating Metabolites and the Intestinal Microbiome
Brief Title: Identifying Periods of High Training Load Considering the Menstrual Cycle Phases in Elite and Non-elite Female Athletes
Status: Recruiting | Type: Observational
Sponsor: Wingate Institute (Other)
Collaborators: Weizmann Institute of Science (Other); Kaplan Medical Center (Other); Ministry of Innovation, Science and Technology of Israel (Unknown)
Responsible Party: Sponsor
Other Study IDs: MC study
Record Dates: First submitted 2024-01-31; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-01

CONDITIONS: Menstrual Cycle; Athletes; Physical Activity
Keywords: Menstrual cycle; Training load; Microbiome; Elite athletes
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Regular cycle: Regular cycle length between 21-35 days.
  Interventions: Behavioral: Effect of training loads and sport performance level on health and sport performance
- Irregular/contraceptives: Irregular cycles (under 21 days or more than 35 days). Contraceptives use of any type (Hormonal intervention).
  Interventions: Behavioral: Effect of training loads and sport performance level on health and sport performance

INTERVENTIONS:
Behavioral: Effect of training loads and sport performance level on health and sport performance — Effect of training loads and sport performance level on health and sport performance

SUMMARY:
Despite a rise in the number of women participating in competitive sports, there remains a gender gap within sport and exercise science literature. Studying females involves potential "noise" through the change in hormone concentrations during the different phases of the female menstrual cycle (MC) which can potentially affect physiological parameters, thereby making study design and interpretation of findings difficult. Longitudinal data on the acute and chronic combined effects of training load and MC phases on circulating female hormones in elite and non-elite female athletes is lacking.

The investigators aim to characterize and track the potential effects of training load and MC phases on performance, anthropometric measures, sport emotions, intestinal microbiome, serum metabolites and injury prevalence in elite and non-elite female athletes.

200 competitive premenopausal female athletes will be recruited. In a longitudinal observational design, each participant will be followed for 1 year, and tested at three time points. At each point, data will be collected on two occasions reflecting distinct phases of the MC.

Finding the possible relationship between the MC phases, training load and performance or specific bio-markers for training load are of utmost importance and can assist professionals to identify periods of high load and over-training, thus preventing injuries and training adjustment.

DETAILED DESCRIPTION:
The purpose of the current investigation is threefold:

1. To evaluate the prevalence of menstruation and menstrual related issues among elite and non-elite female athletes.
2. To identify physical- and bio-markers holding information about training load among elite and non-elite female athletes, using sets of performance measures, hormonal responses, metabolites in the blood and intestinal microbiome
3. To track and characterize the association of training load with a variety of performance (e.g., force, flexibility, endurance etc) and anthropometric measures, sports emotions and affect, rate of perceived exertion (RPE), and injury prevalence in women with different training status (elite and non-elite).

Methods Participants will be tested at three distinct time points that will reflect the different training loads (low, moderate, high) during a year of follow up.

Elite athletes will be tested at: 1. low load phase (baseline); 2. Moderate (training phase prior to competition); 3. High (after training camps or during competitions period).

Testing for each phase will be scheduled for at least two weeks after the beginning of the phase and/or when at least 50% of the duration of the phase is completed. This is to allow for accumulation of training load and phase fatigue or recovery.

Since non elite athletes usually do not follow a periodized training program they will be tested at three time points during the year. The Investigators will similarly aim that these time points will reflect different training loads (low, moderate, and high).

Study description Elite athletes will be recruited through elite athletes' coaches and unions and advertisement using flyers and social media. Non-elite athlete will be recruited through advertisements at Wingate institute and social media.

They will be asked to arrive to a meeting at Wingate institute in which they will receive an explanation about the study by the authorized physician and will sign an informed consent form.

After enrollment, each athlete in the elite group (and coach in the case of an athlete that is part of a team) and non-elite group will meet with one of the investigators to go over their yearly training plan to characterize past and present training history and to establish training phases and schedule individual testing sessions.

The menstrual status of each athlete will be considered when designing the testing schedule, (see blood tests below).

During each of the three assessment periods (low, moderate, high), the athletes will perform the following tests mentioned in study procedures. The Study procedures will be done in addition to the routine follow-up of each athlete.

Study procedures Questionnaires

Participants will be asked to fill the following questionnaires:

Questionnaire 1 -medical history, women health, and physical activity Questionnaire 2- Food frequency Questionnaire (FFQ) Questionnaire 3- Psychological aspects of competition Questionnaire 4- A wellness questionnaire to be filled on each Training load quantification.

Each questionnaire will be filled three times yearly at each of the designated three time periods. The questionnaires will be filled via specific online app designated for research purposes.

Menstrual records During the 12-month period, subjects will be instructed to keep a menstrual calendar using a designated smartphone application to estimate the length of the cycle. They will be asked to record the date of the menses, length of menses, severity of blood flow and any discomfort if it exists.

Blood tests will be drawn by authorized and trained study personal between 8:00 - 10:00 AM after an 8-hour fast, 3 hours of awakens and without any morning training that day. Participants will be asked to avoid taking any medications at the morning of the tests and any supplements three days before the tests.

The blood parameters that will be evaluated are the following: 25OHD, albumin, cortisol, insulin, glucose, TSH, FT4, FT3, total testosterone, testosterone free, SHBG, GH, IGF1. In addition, two aliquots of serum will be frozen for future potential analysis. An additional chemistry tube will be taken for serum metabolites to be analyzed at the Elinav Lab (see below).

Tubes will be centrifuged, and serum/plasma will be frozen at -20 degrees until further analysis at a certified Lab and the Elinav Lab.

The following schedule for blood tests will be employed:

In athletes reporting regular cycles: blood tests will be performed during the follicular phase in days 3-5 of the cycle and again during the luteal phase during days 21-22. These time points were chosen since they represent two occasions where hormones contrast at their greatest magnitude. Participants will alert the researchers on the first day of bleeding and then the 1st session of testing will occur within 3-5 days.

In athletes reporting menses intervals above 35 days or less than nine menstrual cycles per year or if data is unknown - blood tests will be performed three times a year during the different training phases.

Likewise, blood tests will be performed in regular intervals for those athletes using oral contraceptives.

Targeted and untargeted serum metabolomics An untargeted high-performance liquid-chromatography mass-spectrometry is used to characterize the small molecules profile in fecal/plasma samples (i.e. metabolomics). This method identifies different small molecules in a homogenized tissue lysate by simultaneously assessing their molecular weight and electrical charge. In short, a tissue extract is divided into five fractions: one is saved as backup and the rest are analyzed in 4 protocols to identify polar, semi-polar, lipid, and volatile metabolites. Signals are mapped to a known metabolomic database, filtered to optimize signal-to-noise ratio, and normalized. Analysis of clustering and differential abundance then follow to identify candidate key-metabolites that may be correlate with the disease/condition.

Stool microbiome Participants will receive kits in order to collect stool samples at home, and store it in their home freezers until they will be delivered to the Elinav lab at the Weizmann Institute, where they will be stored encoded at -80C, with no identifying information and examined later on.

For microbiome characterization, the investigators will perform whole-genome shotgun metagenomics sequencing, a technique that enables sampling all genes in all organisms present in each sample, including unknown unculturable bacteria. Genetic material is purified from a human microbiome sample and broken down to short fragments that can be sequenced on a large scale in parallel. By comparing these sequences to databases of known microbial genomes, The investigators can characterize the microbial diversity of the sample (which bacteria are present and their abundances, including high-resolution identification of distinct bacterial strains). Using gene abundances, The investigators can reconstruct metabolic pathways and describe the functional capacities of the microbial community that potentially contribute to the phenotype of interest.

Performance Testing procedures Performance measures, covering a broad array of general physical abilities, will include the following tests: maximal aerobic capacity - VO2max test; explosive power - countermovement jump (CMJ); flexibility - sit and reach and ankle dorsiflexion range of motion; strength - maximal voluntary isometric hand grip test (IGT) and isokinetic strength during knee extension (KE) and flexion (KF); and kinematic analysis of frontal plane projection angle (FPPA) as a measure of knee valgus.

Injury Monitoring The investigators will record the prevalence of injuries sustained during the study. Injuries will be documented according to the International Olympic Committee consensus guidelines. Injuries will be classified according to onset, severity, mechanism of injury, body area injured and diagnosis of injury. An injury surveillance questionnaire will be completed by the relevant medical professional working with the athletes as part of the routine follow-up of the athletes.

Training load quantification and wellness The athletes will be instructed to report all their training and competitions during the duration of the study. Endurance athletes will be encouraged to use a Garmin watch , and an online training monitoring interface, TrainingPeaks or Garmin Connect . Acute training load (ATL) will be calculated as the load during the 7 days preceding each assessment date, both as accumulated and average training hours, intensity levels (% time in different training zones), and possibly total and average power or distance covered based on the athlete's individual sport. Chronic training load (CTL) will be defined as the accumulated load for the 4 weeks preceding each assessment date.

In sports in which no objective measurable data exists (e.g., team sports, combat sports etc.), the internal load will be quantified based on the session RPE (sRPE) and the athlete will be asked to keep a training diary and report their training sessions. At the end of each training session the athletes will be asked to subjectively rate the intensity of the entire training session using the category Borg scale (CR-10). The RPE value will then be multiplied by the total duration (min) of the training session. In the non-elite group, the athletes will be encouraged to keep a training diary and report their training duration, distance, type of training and rate the intensity of the training session based on the Borg scale.

The participants will be asked to fill a Wellness status using a subjective wellness questionnaire. The questionnaire is composed of 6 questions evaluating athlete's fatigue, stress, sleep quality, muscle soreness, illness and desire to train on a 7-point scale (1: very, very bad; 7: very, very good). The participants will be asked to fill the questionnaire on a daily basis 2-3 weeks preceding each assessment date.

Anthropometric measures will be done at each of the designated time periods: Height (cm) and body mass (kg) will be measured using a stadiometer and a digital scale respectively, and will be recorded to the nearest 0.1 cm and 0.1 kg, respectively. Body composition [% body fat and lean body mass (kg)] will be evaluated using Dual-Energy X-ray Absorptiometry (DEXA).

Food intake diary - energy availability On top of the FFQ, athletes will receive a detailed explanation on how to record a daily food diary from the investigators. "Energy availability" will be defined as the amount of dietary energy remaining for other bodily functions after exercise training. Dietary energy will be calculated in each subject from a prospective 3-day food diary prior to each assessment session using a Nutrient Analysis program. All subjects will meet with the same registered dietitian and explanations will be given on how to complete the intake (e.g., portion sizes and ounces of liquid consumed). Subjects will be encouraged to weigh portion sizes. "Energy expenditure" will be calculated from duration of sports participation, intensity of exercise, weight, age and sex from the Ainsworth compendium of physical activity. Energy availability will be expressed as kcal/kg lean body mass. energy balance will be considered > 45 kcal·kg-1 FFM·d-1 in healthy young women, and low energy availability will be defined as energy availability <45 kcal/LBM. If the dietitian will realize that the food diary completed by the participant is not reliable or data is missing, a 24hr food and hydration recall will be completed.

Psychological parameters: Emotions and affect. Participants will be asked to a questionnaire which will measure their general affect and their specific emotions related to a specific event and precompetitive emotion. Two primary general dimensions of mood, positive and negative affect, will be measured by using the Positive-Affect Negative-Affect Scale and the Sport Emotion Questionnaire is a sport-specific measure of precompetitive emotion grounded in the experience of athletes, assessing: anger, anxiety, dejection, excitement, and happiness.

ELIGIBILITY:
Inclusion Criteria:

* Elite athletes are defined as participating and competing at national and/or international level at their sports.
* Non-elite athletes are defined as performing at least 3 hours of physical activity per week.

Exclusion Criteria:

* Currently pregnant or lactating or planning a pregnancy in the following year.
* Regular drug use which may affect performance, including but not limited to performance enhancing drugs.
* Any medical diagnosis, including recent or current injury, which could affect performance and/or health under the discretion of the study team.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biologically female
Study Population: Competitive elite and non-elite female athletes.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Stool Microbiome | 3-6 times during 12 months
  Participants will receive kits in order to collect stool samples at home, and store it in their home freezers until they will be delivered to the Elinav lab at the Weizmann Institute, where they will be stored encoded at -80C. A whole-genome shotgun metagenomics sequencing will be performed on the samples. This will enable the investigators to sample all genes in all organisms present in each sample, including unknown unculturable bacteria.
Serum metabolomics | 3-6 times during 12 months
  An untargeted high-performance liquid-chromatography mass-spectrometry is used to characterize the small molecules profile in plasma samplesץ
VO2max | 3-6 times during 12 months
  Maximal Aerobic power
Countermovement jump | 3-6 times during 12 months
  Countermovement jump performance will be measured using the Optojump Next system. The participants will be instructed to start from an upright position and to descend to a self-selected depth by bending at the hips and knees, immediately followed by a maximal vertical jump effort. Participants' hands will be kept on their hips throughout the entire movement. Participants will perform three attempts, separated by 30 seconds rest. Jump height will be recorded to the nearest 0.1 cm. The best and calculation of average jumps' height will be selected for statistical analysis.
Flexibility | 3-6 times during 12 months
  Sit and reach and ankle dorsiflexion range of motion
Grip Strength | 3-6 times during 12 months
  Maximal voluntary isometric hand grip
Lower leg Strength | 3-6 times during 12 months
  Isokinetic strength during Knee extension and flexion
Blood tests | 3-6 times during 12 months
  Blood tests will draw in the morning in a fasted state. The following parameters will be evaluated from the plasma: TSH (mlU/l), FT4 (pmol/l), FT3 (pmol/l), GH (ng/ml), IGF-1 (nmol/l), Testosterone total (nmol/l), Testo free (nmol/l), SHBG (nmol/l), Insulin (mU/l), 25OHD (nmol/l), Albumin (g/dl), Cortisol (nmol/l), Glucose (mg/dl)
Knee valgus | 3-6 times during 12 months
  This test assesses dynamic knee valgus during a double leg drop jump using the reliable method of calculating the frontal plane projection angle. The athlete will perform a drop jump from a 30cm box landing with each foot on a force plate then immediately exploding upwards into a vertical jump. The athlete will be videoed using a video camera placed directly in front of the subject, 5m away. Markers will be placed by an experienced clinician on the midpoint of the femoral condyles, midpoint of the ankle malleoli, and proximal thigh along a line from the ASIS to the knee marker. The angle between line from the proximal thigh to the knee joint and line from the knee joint to the ankle at maximum knee flexion. Knee valgus = positive angle; Knee varus = negative angle. Reactive strength index will be calculated from force plate data providing information on plyometric performance, reactive jump capacity and dynamic explosive ability. The athlete will perform two drop jumps.

SECONDARY OUTCOMES:
Anthropometric (Height) | 3-6 times during 12 months
  Height in centimeters
Psychological questionnaire (Positive-Affect Negative-Affect scale - PANAS) | 3-6 times during 12 months
  Two primary general dimensions of mood, positive and negative affect, will be measured by using the Positive-Affect Negative-Affect Scale. The 20-items scale is internally consistent and has excellent convergent and discriminant correlations with lengthier measures of the same underlying mood factors. The participants will be asked to rate themselves on a five-point Likert scale.
Anthropometric (Weight) | 3-6 times during 12 months
  Body mass in kg
Percentage body fat (%) | 3-6 times during 12 months
  Body fat will assessed using Dexa

OTHER OUTCOMES:
Psychological questionnaire (The Sport Emotion Questionnaire (SEQ) | 3-6 times during 12 months
  The Sport Emotion Questionnaire (SEQ) is a sport-specific measure of precompetitive emotion grounded in the experience of athletes, assessing: anger, anxiety, dejection, excitement, and happiness. The SEQ shows good evidence of validity and reliability and represents a range of emotions with greater emphasis on positive emotions than that provided by other available group-oriented measures for use in sport research. The participants will be asked to rate themselves on a five-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Rotem Kislev-Cohen, Ph.D, Principal Investigator — Wingate Institute
Locations (1):
- Wingate Institute, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sims ST, Heather AK. Myths and Methodologies: Reducing scientific design ambiguity in studies comparing sexes and/or menstrual cycle phases. Exp Physiol. 2018 Oct;103(10):1309-1317. doi: 10.1113/EP086797. Epub 2018 Aug 15. PMID 30051938
- [Background] Pallavi LC, D Souza UJ, Shivaprakash G. Assessment of Musculoskeletal Strength and Levels of Fatigue during Different Phases of Menstrual Cycle in Young Adults. J Clin Diagn Res. 2017 Feb;11(2):CC11-CC13. doi: 10.7860/JCDR/2017/24316.9408. Epub 2017 Feb 1. PMID 28384857
- [Background] Bahr R, Clarsen B, Derman W, Dvorak J, Emery CA, Finch CF, Hagglund M, Junge A, Kemp S, Khan KM, Marshall SW, Meeuwisse W, Mountjoy M, Orchard JW, Pluim B, Quarrie KL, Reider B, Schwellnus M, Soligard T, Stokes KA, Timpka T, Verhagen E, Bindra A, Budgett R, Engebretsen L, Erdener U, Chamari K. International Olympic Committee consensus statement: methods for recording and reporting of epidemiological data on injury and illness in sport 2020 (including STROBE Extension for Sport Injury and Illness Surveillance (STROBE-SIIS)). Br J Sports Med. 2020 Apr;54(7):372-389. doi: 10.1136/bjsports-2019-101969. Epub 2020 Feb 18. PMID 32071062
- [Background] Nattiv A, Loucks AB, Manore MM, Sanborn CF, Sundgot-Borgen J, Warren MP; American College of Sports Medicine. American College of Sports Medicine position stand. The female athlete triad. Med Sci Sports Exerc. 2007 Oct;39(10):1867-82. doi: 10.1249/mss.0b013e318149f111. PMID 17909417
- [Background] Ainsworth BE, Haskell WL, Whitt MC, Irwin ML, Swartz AM, Strath SJ, O'Brien WL, Bassett DR Jr, Schmitz KH, Emplaincourt PO, Jacobs DR Jr, Leon AS. Compendium of physical activities: an update of activity codes and MET intensities. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S498-504. doi: 10.1097/00005768-200009001-00009. PMID 10993420
- [Background] Ashley CD, Kramer ML, Bishop P. Estrogen and substrate metabolism: a review of contradictory research. Sports Med. 2000 Apr;29(4):221-7. doi: 10.2165/00007256-200029040-00001. PMID 10783898
- [Background] D'Eon TM, Sharoff C, Chipkin SR, Grow D, Ruby BC, Braun B. Regulation of exercise carbohydrate metabolism by estrogen and progesterone in women. Am J Physiol Endocrinol Metab. 2002 Nov;283(5):E1046-55. doi: 10.1152/ajpendo.00271.2002. PMID 12376334
- [Background] Elliott-Sale KJ, Minahan CL, de Jonge XAKJ, Ackerman KE, Sipila S, Constantini NW, Lebrun CM, Hackney AC. Methodological Considerations for Studies in Sport and Exercise Science with Women as Participants: A Working Guide for Standards of Practice for Research on Women. Sports Med. 2021 May;51(5):843-861. doi: 10.1007/s40279-021-01435-8. Epub 2021 Mar 16. PMID 33725341